CLINICAL TRIAL: NCT00773370
Title: Adaptive Physical Activity for Chronic Stroke
Acronym: APA-Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Maryland, Baltimore County (Other); Howard County Office on Aging (Unknown); MedStar National Rehabilitation Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B6329-R; H 30467 (Other: UMB BRAAN Number); HP-00044066 (Other: UMB CICERO Number)
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Stroke
Keywords: stroke; exercise
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APA-Stroke (Experimental): The APA-stroke exercise program designed specifically for individuals with hemiparetic gait deficits due to stroke. These progressive exercises focus on walking, balance and weight shifting and include an exercise homework component.
  Interventions: Behavioral: APA-Stroke
- Sittercise (Active Comparator): Sittercise is not stroke specific. This less vigorous exercise program consists of seated exercise, focusing on stretching to improve general range of motion and weight exercises to strengthen the trunk, arms, and legs. There is no assigned exercise homework associated with this group.
  Interventions: Behavioral: Sittercise

INTERVENTIONS:
Behavioral: APA-Stroke — Exercise program design specifically for individuals with residual hemiparetic gait deficits due to stroke. Exercises are progressive, beginning with a 5 minute walk at the beginning and end of each class and gradually progressing to a 15 minute walk at the beginning and end of each class. Exercises focus on walking and are designed to improve walking ability and balance. Program includes a homework component.
  Arms: APA-Stroke
Behavioral: Sittercise — Not stroke specific. This less vigorous exercise program consists of seated exercise focusing on stretching to improve general range of movement and weight exercises to strengthen the trunk, arms, and legs. There is no assigned exercise homework.
  Arms: Sittercise

SUMMARY:
This study will compare the Adaptive Physical Activity program (APA) to a less vigorous group exercise program, (Sittercise) to see if APA leads to greater improvements in walking endurance, quality of life, and participation in social activities.

DETAILED DESCRIPTION:
The purpose of this study is to translate the Italian APA exercise model into a sustainable, evidence-based VA community program of exercise for older adults with chronic stroke. The investigators' short-term objectives are to test study hypotheses using a Randomized Clinical Trial (RCT) with an Attention Control (also referred to as the "Sittercise" exercise program). The investigators will also explore factors related to exercise adherence in a community program for chronic stroke survivors. The investigators' longer term objective is to disseminate this model to facilitate the development of a network of community-based exercise programs for older adults with chronic stroke. In the RCT the investigators propose to offer courses in Office of Aging (OoA) Senior Centers and National Rehabilitation Hospital. At the conclusion of the research study, the OoA plans to continue offering APA-stroke courses. Through partnership, the Veterans Health Administration (VHA) and the Administration of Aging (AoA) can potentially replicate this model at the community throughout the U.S. using local OoA Senior Centers and other facilities that would increase community access for Veterans.

ELIGIBILITY:
Inclusion Criteria:

* evidence of stroke (ischemic or hemorrhagic) minimum 6 months prior in men or women ages 40 or older;
* residual hemiparetic gait deficits;
* already completed all conventional inpatient and outpatient physical therapy;
* ability to rise from a chair unaided and without an assistive device

Exclusion Criteria:

* cardiac history of active unstable angina, recent (less than 3 months) myocardial infarction, or congestive heart failure (NYHA category II or higher);
* orthopedic, circulatory, or chronic pain conditions restricting exercise;
* active cancer; poorly controlled hypertension ( greater than 180/100 on 2 readings separated by 5 minutes rest);
* dementia;
* severe receptive or global aphasia with inability to follow 2-step commands;
* co-morbid non-stroke neurological disorder that impairs mobility (e.g. multiple sclerosis or Parkinson's);
* untreated clinical depression;
* inability to complete the "6-Minute Walk" test during baseline testing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-01; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Stuart, ScD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (2):
- United States (2):
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | APA-Stroke | Sittercise
Started | 43 | 33
Completed | 25 | 23
Not Completed | 18 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APA-Stroke | Sittercise | Total
Number analyzed (Participants) | 43 | 33 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.2) | 65 (11.7) | 64 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 22 | 17 | 39
Race/Ethnicity, Customized [Number; unit: participants]
  White | 17 | 13 | 30
  Black | 24 | 14 | 38
  Other | 1 | 6 | 7
  Missing | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 43 | 33 | 76
Hemiparesis [Number; unit: participants]
  Left | 27 | 18 | 45
  Right | 13 | 13 | 26
  Missing | 3 | 2 | 5
Year since stroke [Mean (Standard Deviation); unit: years] | 5.5 (5.2) | 4.7 (8.5) | 5.2 (6.6)
Berg Balance [Mean (Standard Deviation); unit: units on a scale] — The Berg consists of 14 items, each graded on a scale of 0-4. A score for the Berg could in theory range from a minimum of 0 to a maximum of 56. A score below 45 is indicative of balance impairment; thus the lower the score the greater the fall risk.
  units on a scale | 44.76 (9.03) | 43.00 (9.02) | 44.58 (9.03)
Short Physical Performance Battery (SPPB) [Mean (Standard Deviation); unit: units on a scale] — Components include gait speed, a repeated chair stand, and a standing balance test. Scores for gait speed, chair stand, and total balance are calculated and then summed for the total score. Each component can range from 0-4 points, thus the maximum composite score can range from 0-12 points, with 0 reflecting the lowest functioning while a score of 12 indicates the subject reached the maximum measured competency in all three domains.
  units on a scale | 6.60 (2.66) | 6.06 (2.64) | 6.36 (2.65)
6 Minute Walk Test (MWT) [Mean (Standard Deviation); unit: meters] | 189.07 (97.38) | 171.69 (97.42) | 181.52 (97.40)
Stroke Impact Scale (SIS) [Mean (Standard Deviation); unit: units on a scale] — SIS Version 3.0 is a self report scale that includes 59 items and assesses 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, and participation/role function). Summative scores for each domain range from 0-100. Total scores range from 0-800. A higher score reflects better function.
  units on a scale | 466.62 (201.75) | 490.79 (201.76) | 476.29 (201.75)

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Test (6MWT)
Description: Total distance walked for 6 minutes (in meters) is the primary outcome measure. Participants use the same assistive devices and/or orthoses they use when walking across a parking lot. They are instructed to cover as much distance as they can over a flat 100 foot walking surface demarcated by traffic cones during the six minute time period. Change in distance covered is the outcome variable of interest for this study. Walking a greater distance (e.g. more meters during the 6 minute test) reflects improvement in walking speed and endurance. We computed the slopes (i.e. rates of change from baseline to 3-months and 6-months) using a random effects ANOVA (random intercept and random slope), and determined if the slopes were different using unpaired Student's t-tests.
Time Frame: measured at baseline, 3 months, 6 months
Measure: Mean (Standard Error); unit: meters
Arm/Group | APA-Stroke | Sittercise
Number analyzed (Participants) | 25 | 23
meters
  Baseline | 189 (15) | 172 (17)
  Three-months | 211 (21) | 170 (23)
  Six-Months | 228 (22) | 167 (23)
Statistical Analysis 1: Comparison: APA-Stroke vs Sittercise; Test type: Superiority or Other; p < 0.25, ANOVA — Random effects ANOVA with random intercept and random slope compared the time course (slopes) of change in our outcome measures across three time points: baseline, three, and six-months in our two experimental groups--APA-stroke and Sittercise; difference between slopes = 8.43, Standard Deviation 7.17
Statistical Analysis 2: Comparison: APA-Stroke; Within group change over time; Test type: Superiority or Other; p < 0.004, ANOVA — Random effects ANOVA, random intercept, random slope estimating within group change (slope) over time; Slope = 14.95, Standard Deviation 4.92
Statistical Analysis 3: Comparison: Sittercise; Within group change over time; Test type: Superiority or Other; p = .218, ANOVA — Random effects ANOVA, random intercept, random slope estimating within group change (slope) over time; Slope = 6.52, Standard Deviation 5.13

2. Secondary Outcome: Balance as Measured by the Berg Balance Scale (BBS)
Description: The Berg is a widely used test for assessing balance and to predict fall risk in the elderly. It has been validated with patients post stroke. The Berg consists of 14 items, each graded on a scale of 0-4. Thus a score for the Berg could in theory range from a minimum of 0 to a maximum of 56. A score below 45 is indicative of balance impairment; thus the lower the score the greater the fall risk. We computed the slopes (i.e. rates of change from baseline to 3-months and 6-months) using a random effects ANOVA (random intercept and random slope), and determined if the slopes were different using unpaired Student's t-tests.
Time Frame: measured at baseline, 3 months, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | APA-Stroke | Sittercise
Number analyzed (Participants) | 25 | 23
units on a scale
  Baseline | 44.8 (1.1) | 43.0 (1.9)
  Three-Months | 46.5 (1.5) | 43.0 (2.0)
  Six-Months | 47.6 (1.1) | 41.6 (2.3)
Statistical Analysis 1: Comparison: APA-Stroke vs Sittercise; Test type: Superiority or Other; p = .47, ANOVA — [p-value comment as in outcome 1, analysis 1]; Difference between slopes = 0.186, Standard Deviation 0.256
Statistical Analysis 2: Comparison: APA-Stroke; Within group change over time; Test type: Superiority or Other; p = .225, ANOVA — Random effects ANOVA, random intercept, random slope estimating within group change (slope) over time; Slope = .215, Standard Deviation 0.175
Statistical Analysis 3: Comparison: Sittercise; Within group change over time; Test type: Superiority or Other; p = .88, ANOVA — Random effects ANOVA, random intercept, random slope estimating within group change (slope) over time; Slope = .029, Standard Deviation 0.187

3. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: The SPPB, which is extensively used in stroke studies, includes three components and a composite score. Components include gait speed, a repeated chair stand, and a standing balance test. Scores for gait speed, chair stand, and total balance are calculated and then summed for the total score. Each component can range from 0-4 points, thus the maximum composite score can range from 0-12 points, with 0 reflecting the lowest functioning while a score of 12 indicates the subject reached the maximum measured competency in all three domains. We computed the slopes (i.e. rates of change from baseline to 3-months and 6-months) using a random effects ANOVA (random intercept and random slope), and determined if the slopes were different using unpaired Student's t-tests.
Time Frame: measured at baseline, 3 months, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | APA-Stroke | Sittercise
Number analyzed (Participants) | 25 | 23
units on a scale
  Baseline | 6.60 (.40) | 6.10 (.48)
  Three-Months | 6.76 (.48) | 5.92 (.50)
  Six-Months | 7.12 (.51) | 5.96 (.61)
Statistical Analysis 1: Comparison: APA-Stroke vs Sittercise; Test type: Superiority or Other; p = .98, ANOVA — [p-value comment as in outcome 1, analysis 1]; Difference between slopes = .002, Standard Deviation .078
Statistical Analysis 2: Comparison: APA-Stroke; Within group change over time; Test type: Superiority or Other; p = .54, ANOVA — Random effects ANOVA, random intercept, random slope estimating within group change (slope) over time; Slope = .033, Standard Deviation .054
Statistical Analysis 3: Comparison: Sittercise; Within group change over time; Test type: Superiority or Other; p = .59, ANOVA — Random effects ANOVA, random intercept, random slope estimating within group change (slope) over time; Slope = .031, Standard Deviation 0.057

4. Secondary Outcome: Stroke Impact Scale (SIS)
Description: The SIS Version 3.0 is a self report scale widely used to assess health status after stroke. It includes 59 items and assesses 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, and participation/role function). The SIS uses a 5-point Likert Scale. Summative scores for each domain range from 0-100. Total scores range from 0 to 800. A higher score reflects better function. We computed the slopes (i.e. rates of change from baseline to 3-months and 6-months) using a random effects ANOVA (random intercept and random slope), and determined if the slopes were different using unpaired Student's t-tests.
Time Frame: measured at baseline, 3 months, 6 months
Population: SIS data were incomplete for six sittercise participants, hence the discrepancy between number of participants analyzed and the flow data reported above.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | APA-Stroke | Sittercise
Number analyzed (Participants) | 25 | 17
units on a scale
  Baseline | 467 (32) | 491 (36)
  Three-Months | 463 (35) | 576 (17)
  Six-Months | 562 (23) | 579 (18)
Statistical Analysis 1: Comparison: APA-Stroke vs Sittercise; Random effects ANOVA with random intercept and random slope was used to compare the time course of change in our outcome measures across three time points: baseline, three, and six-months in our two experimental groups--APA-stroke and Sittercise; Test type: Superiority or Other; p = .98, ANOVA; Slope = 0.296, Standard Deviation 9.77
Statistical Analysis 2: Comparison: APA-Stroke; Test type: Superiority or Other; p = .02, ANOVA — Random effects ANOVA, random intercept, random slope estimating within group change (slope) over time; Slope = 15.49, Standard Deviation 6.19
Statistical Analysis 3: Comparison: Sittercise; Test type: Superiority or Other; p = .051, ANOVA — Random effects ANOVA, random intercept, random slope estimating within group change (slope) over time; Slope = 15.193, Standard Deviation 7.553

ADVERSE EVENTS:
Arm/Group | APA-Stroke | Sittercise
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/33
Other Adverse Events (participants affected / at risk) | 6/43 | 4/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APA-Stroke (N=43) | Sittercise (N=33)
muscle pain (Musculoskeletal and connective tissue disorders) | 1 | 2
faintness (Cardiac disorders) | 2 | 0
fall (Musculoskeletal and connective tissue disorders) | 1 | 2 — Controlled fall without injury
shortness of breath (Cardiac disorders) | 1 | 0
chest pain (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No